CLINICAL TRIAL: NCT01531452
Title: a Phase II Study of Oxaliplatin Plus S-1 (SOX) as First-line Treatment for Patients With Advanced Gastric Cancer
Brief Title: The Efficacy of Oxaliplatin Plus S-1 for Treatment of Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Lin Yang, MD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-016
Record Dates: First submitted 2012-02-06; First posted 2012-02-13 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; drug therapy; oxaliplatin; s1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment (Experimental): oxaliplatin+s1
  Interventions: Drug: Oxaliplatin; Drug: s1

INTERVENTIONS:
Drug: Oxaliplatin — 130mg/m2 d1,repeated q21d
  Other Names: eloxatin
Drug: s1 — 80mg/m2/d, d1-14,repeated q21d
  Other Names: TS-1

SUMMARY:
The purpose of this study is to determine the efficacy and safety of oxaliplatin and s1 as first-line treatment of advanced gastric cancer.

DETAILED DESCRIPTION:
There was no evidence of standard chemotherapy for advanced gastric cancer (AGC) in China. Fluoropyrimidines and cisplatin have been widely used in a variety of combinations in the treatment of AGC. Capecitabine/cisplatin combination therapy showed an overall response rate (ORR) of 41- 55%, a median time to progression/progression free survival (TTP/PFS) of 5.6-6.3 months, and a median overall survival (OS) of 10.1-10.5 months. Though no studies have compared two oral fluoropyrimidines in combination with oxaliplatin, both S-1 and capecitabine appear to be comparable in terms of efficacy and safety. The investigators conducted a phase II trial of oxaliplatin combined with S-1 in the treatment of first-line AGC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven in operable advanced gastric adenocarcinoma (including adenocarcinoma of the gastrooesophageal junction) or relapse gastric adenocarcinoma
* Measurable lesion and/or non-measurable lesion defined by RECIST
* ECOG performance status ≦ 1
* Hgb ≧ 8g/dL, WBC 4000-12000/mm3, platelets ≧ 100,000/mm3
* Creatine ≦ upper normal limit (UNL)
* Total bilirubin ≦ 1.5 X UNL
* AST, ALT and ALP ≦ 2.5 x UNL
* Subjects must be able to take orally
* No prior chemotherapy
* Life expectancy estimated than 3 months
* Written informed consent

Exclusion Criteria:

* Pregnancy or lactation women, or women with suspected pregnancy or men with willing to get pregnant
* Known brain metastases
* History of hypersensitivity to fluoropyrimidines, oxaliplatin
* Active double cancer
* Treatment with any investigational product during the last 4 weeks prior to study entry
* Symptomatic peripheral neuropathy ≧ garde 2. by NCI-CTCAE ver.3.0
* Any previous chemotherapy or radiotherapy for AGC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-06; Primary Completion 2012-11 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 2 years
  from date of treatment was administered until the date of first documented progression or death from any cause whichever first, assessed every 6 weeks

SECONDARY OUTCOMES:
Response Rate | 2 years
  From date of treatment was administered until the date of first documented response to treatment according to RECIST criteria,assessed every 2 cycles
overall survival | 2 years
  From date of treatment was administered until the date of death from any cause,assessed every 3 months
number of participants with adverse events | 2 years
  assessed from treatment was administered until 1 months after withdrawing from study

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, MD, Principal Investigator — cancer hospital&institute,Chinese Academy of Medical Sciences
Locations (1):
- cancer hospital & Institute,Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China